CLINICAL TRIAL: NCT06933836
Title: How Does First Line Treatment With DSLT Perform in Treatment-naïve Patients With Newly Diagnosed Primary Open Angle Glaucoma
Brief Title: DSLT Performance in Treatment-naïve Patients With Newly Diagnosed Open Angle Glaucoma
Status: Recruiting | Type: Observational
Sponsor: Barnet Dulaney Perkins Eye Centers (Network)
Collaborators: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Alcon - IIT Proposal 95645649
Record Dates: First submitted 2025-03-04; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Open Angle Glaucoma (OAG)
Keywords: Glaucoma; DSLT; Interocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment naïve (including medication in either eye, previous laser or surgery) mild to moderate POA: (including medication in either eye, previous laser or surgery) mild to moderate POA
  Interventions: Device: DSLT enables newly diagnosed patients to remain well controlled and off medications

INTERVENTIONS:
Device: DSLT enables newly diagnosed patients to remain well controlled and off medications — DSLT enables newly diagnosed patients to remain well controlled and off medications

SUMMARY:
DSLT demonstrates a ≥ 20% reduction of IOP from pre-treatment baseline in POAG patients naïve of previous glaucoma treatment at 12 months.

DETAILED DESCRIPTION:
DSLT enables newly diagnosed patients to remain well controlled and off medications

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Patients age 30 or greater with an IOP of 18-26 mmHg
* Mild to moderate POAG patients (mild or moderate according to the AAO PPP Guidelines)
* DSLT procedure

Exclusion Criteria:

* History of prior glaucoma treatment - this includes past medication use (in either eye), previous lasers or incisional surgery
* Angle closure patients
* Ocular Hypertension
* Baseline VF MD of worse than -12dB
* Uncontrolled systemic microvascular disease (eg. HTN, DM)
* Subjects with peri-limbal findings (e.g. melanosis, tumors, extensive pterygium, significant senile arcus and pterygium)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 55 Treatment naïve (including medication in either eye, previous laser or surgery) mild to moderate POAG subjects
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Success of IOP Reduction Through DSLT Utilization | 12 months
  Proportion of patients (%) with DSLT success as defined as IOP lowering of >20% and no additional medications or procedures at 12 months.

SECONDARY OUTCOMES:
Other Improvements to Disease State through DSLT Treatment | 12 months
  • Change in mean deviation.. (dB)
Other Improvements to Disease State through DSLT Treatment | 12 months
  • Change in RNFL /GCA (µm)
Other Improvements to Disease State through DSLT Treatment | 12 months
  • Overall IOP reduction (mmHG)
Other Improvements to Disease State through DSLT Treatment | 12 months
  • Medication reduction (#0-5)
Other Improvements to Disease State through DSLT Treatment | 12 months
  • SSIs (% on trabeculectomy, glaucoma drainage implant (GDI), other)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Funke, Medical Doctor, Principal Investigator — Barnet Dulaney Perkins Eye Centers
Locations (1):
- Barnet Dulaney Perkins Eye Centers, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study collection, the investigators will share the findings of the DSLT treatment with other researchers to then be published
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be available after the study is completed tentatively 12/2026 and available for 12 months until 12/2027.
Access Criteria: The investigators will allow other researchers to contact us for information and the study results, the final results is the only thing that others will have access to upon request.
URL: http://goodeyes.com

REFERENCES:
- [Background] Radcliffe N. Direct Selective Laser Trabeculoplasty. Expanding Access to and Delivery of SLT Poses a Great Challenge. Glaucoma Today. 2022.
- [Background] Takusagawa HL, Hoguet A, Sit AJ, Rosdahl JA, Chopra V, Ou Y, Richter G, Kim SJ, WuDunn D. Selective Laser Trabeculoplasty for the Treatment of Glaucoma: A Report by the American Academy of Ophthalmology. Ophthalmology. 2024 Jan;131(1):37-47. doi: 10.1016/j.ophtha.2023.07.029. Epub 2023 Sep 14. PMID 37702635
- [Background] Narayanaswamy A, Leung CK, Istiantoro DV, Perera SA, Ho CL, Nongpiur ME, Baskaran M, Htoon HM, Wong TT, Goh D, Su DH, Belkin M, Aung T. Efficacy of selective laser trabeculoplasty in primary angle-closure glaucoma: a randomized clinical trial. JAMA Ophthalmol. 2015 Feb;133(2):206-12. doi: 10.1001/jamaophthalmol.2014.4893. PMID 25429421
- [Background] Gazzard G, Konstantakopoulou E, Garway-Heath D, Garg A, Vickerstaff V, Hunter R, Ambler G, Bunce C, Wormald R, Nathwani N, Barton K, Rubin G, Buszewicz M; LiGHT Trial Study Group. Selective laser trabeculoplasty versus eye drops for first-line treatment of ocular hypertension and glaucoma (LiGHT): a multicentre randomised controlled trial. Lancet. 2019 Apr 13;393(10180):1505-1516. doi: 10.1016/S0140-6736(18)32213-X. Epub 2019 Mar 9. PMID 30862377
- [Background] Latina MA, Park C. Selective targeting of trabecular meshwork cells: in vitro studies of pulsed and CW laser interactions. Exp Eye Res. 1995 Apr;60(4):359-71. doi: 10.1016/s0014-4835(05)80093-4. PMID 7789416